CLINICAL TRIAL: NCT02227524
Title: Trekking Poles to Aid Multiple Sclerosis Gait Impairment
Acronym: TRAMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rowan University (Other)
Responsible Party: Principal Investigator, Eric Gregory, Director of Research Compliance, Rowan University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: Pro201300052
Record Dates: First submitted 2014-08-20; First posted 2014-08-28 (Estimated); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Walking; Gait
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- No Device (Experimental): Assistive device conditions
  Interventions: Other: No device; Device: Single-point cane (SPC); Device: Four-point cane (FPC); Device: Trekking pole (TP).
- Single Point Cane (Experimental): Assistive device condition
  Interventions: Other: No device; Device: Single-point cane (SPC); Device: Four-point cane (FPC); Device: Trekking pole (TP).
- Four-Point Cane (Experimental): Assistive device condition
  Interventions: Other: No device; Device: Single-point cane (SPC); Device: Four-point cane (FPC); Device: Trekking pole (TP).
- Trekking Pole (Experimental): Assistive device condition
  Interventions: Other: No device; Device: Single-point cane (SPC); Device: Four-point cane (FPC); Device: Trekking pole (TP).

INTERVENTIONS:
Other: No device — Compare walking function and ability in a sample of persons with MS under four different assistive device conditions: no device, single-point cane (SPC), four-point cane (FPC) and trekking pole (TP).
Device: Single-point cane (SPC) — Compare walking function and ability in a sample of persons with MS under four different assistive device conditions: no device, single-point cane (SPC), four-point cane (FPC) and trekking pole (TP).
Device: Four-point cane (FPC) — Compare walking function and ability in a sample of persons with MS under four different assistive device conditions: no device, single-point cane (SPC), four-point cane (FPC) and trekking pole (TP).
Device: Trekking pole (TP). — Compare walking function and ability in a sample of persons with MS under four different assistive device conditions: no device, single-point cane (SPC), four-point cane (FPC) and trekking pole (TP).

SUMMARY:
In this study, the investigators will examine a sample of persons with multiple sclerosis (MS) to determine whether their walking function and ability is different depending on which walking assistive device is used.

DETAILED DESCRIPTION:
In this study, the investigators will examine a sample of persons with multiple sclerosis (MS) to determine whether their walking function and ability is different depending on which walking assistive device is used. In addition, the investigators will examine the psychosocial impact and amount of fatigue induced by each assistive device. Data collection will consist of a series of assessments via survey and physical performance. The analyses will consist of appropriate comparisons of means to determine if the use of different assistive devices alters any of the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Be 18-64 years old with a confirmed diagnosis of MS
* Have perceived walking difficulty
* Have an EDSS score of < 6, calculated by the physician
* Ability to understand study procedures and to comply with them for the entire length of the study

Exclusion Criteria:

* Have had a MS exacerbation in the prior 8 weeks
* Have other serious medical conditions that would impair their ability to participate in gait performance testing (i.e. severe rheumatoid arthritis or osteoarthritis)
* If the physician deems a participant unsafe to go home with devices
* Cannot communicate in English
* Possess greater than a mild decrease in mentation (i.e. a score of >2 on the Mental Functions item of the FSS)
* Inability or unwillingness of individual to give written informed consent

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2014-04; Primary Completion 2019-03-07 (Actual); Study Completion 2019-03-07 (Actual)

PRIMARY OUTCOMES:
Composite measures of walking | 1 year
  Temporal and spatial parameters of gait/walking (measured with the GAITRite portable walkway system)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Barone, DO, Principal Investigator — Rowan University School of Osteopathic Medicine
Locations (1):
- Rowan University School of Osteopathic Medicine, Stratford, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No